CLINICAL TRIAL: NCT00432432
Title: The Efficacy of Combination Methotrexate and Infliximab in Patients With Ankylosing Spondylitis:A Clinical and Magnetic Resonance Imaging Correlation
Brief Title: Combination Methotrexate and Infliximab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS-2005-003
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; MTX; Infliximab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Placebo Comparator): placebo with infliximab
  Interventions: Drug: Infliximab and MTX

INTERVENTIONS:
Drug: Infliximab and MTX — MTX 15mg weekly Infliximab 5mg/kg given at day 0, wk 2, wk6
  Other Names: remicade

SUMMARY:
Combination Methotrexate and Infliximab:Influence of immunogenicity on the efficacy of infliximab in patients with Ankylosing Spondylitis.

DETAILED DESCRIPTION:
Forty consecutive patients will be recruited from the rheumatology clinic of the Prince of Wales Hospital with AS meeting the modified New York criteria with active disease as defined (see below). They will be randomized to receive MTX 7.5 mg/week initially with a weekly 2.5mg increment until 15mg/week dosage is reached,( i.e by week 6) or a placebo together with folic acid 5mg daily for a period of 16 week. After 16 weeks, all patients will receive infliximab at 5 mg/kg per dose, at weeks 16, 18, and 22 (3 doses), and will continue with MTX 15 mg/week or placebo. Thereafter, they will be followed up at week 30, 38 weeks. MRI changes in the sacroiliac joints (SI) before and after infliximab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the AS:meeting the modified New York criteria
* Active disease despite NSAID treatment defined as:
* Spinal inflammation ≧ 30 and a score of 30 on at least two of the other three domains
* Back pain
* Patient global assessment of disease activity
* Physical function
* Informed consent

Exclusion Criteria:

* Complete ankylosis of the spine
* On sulphasalazine
* Previous use of TNF inhibitors
* Multiple use of NSAIDS
* Prednisolone > 10mg/day
* Changes of NSAIDS or dose of prednisolone within 2 weeks of baseline
* Little or no ability for self-care
* Received intra-articular,intramuscular, or intravenous corticosteroids in the 4 weeks before screening
* Infected joint prosthesis during the previous 5 years
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months
* Any chronic infectious disease such as renal infection, chest infection with bronchiectasis or sinusitis
* Active tuberculosis requiring treatment within the previous 3 years
* Opportunistic infections such as herpes zoster within the previous 2 months
* Any evidence of active cytomegalovirus; active Pneumocystis carinii; or drug-resistant atypical mycobacterial infection
* Known hypersensitivity to murine proteins
* Current signs or symptoms of severe,progressive,or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease
* A history of lymphoproliferative disease including lymphoma or signs suggestive of disease, such as lymphadenopathy of unusual size or location (ie,lymph nodes in the posterior triangle or the neck, infraclavicular epitrochlear, or periaortic areas); splenomegaly;
* Any known malignant disease except basal cell carcinoma currently or in the past 5 years.
* A hemoglobin level < 8.5 gm/dl, a white blood cell count < 3.5 × 10^9/liter, a platelet count < 100 × 10^9/liter, a serum creatinine level > 150 µmol/l, serum transaminase levels 1.25 times the upper limit of normal, or alkaline phosphatase levels > 2 times the upper limit of normal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-02; Primary Completion 2006-08 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The number of patient exhibited an ASAS 20 response to treatment at week 20. | wk52

SECONDARY OUTCOMES:
Proportion of patients with 50% and 70% improvement in disease activity.Patient global assessment of disease activity and pain;BASFI;early morning stiffness;physician global assessment of disease activity.Changes in the pre and post infusion MRI. | wk52

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Li, MD, Principal Investigator — Chinese University of Hong Kong